CLINICAL TRIAL: NCT04832685
Title: Neuromodulation of Mind-Wandering in Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Darin Dougherty, MD, Director, Division of Neurotherapeutic, Department of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021P000704
Record Dates: First submitted 2021-03-30; First posted 2021-04-06 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Depression
Keywords: Ultrasound
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Participants will be divided into 2 groups, healthy controls and participants with depression. Both groups will receive sham and active modulation (order counterbalanced).
Masking Description: For sham sonication, a gel pad that absorbs ultrasound will be used with the transducer so that the ultrasound will not go through the skull and into the brain. For active sonication, a gel pad that allows the transmission of ultrasound waves will be used with the transducer. These gel pads look identical; this study will be double-blinded where study staff will not know which gel pad corresponded with active or sham LIFUP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active LIFUP (Active Comparator): All participants will receive active modulation of the posterior cingulate cortex (PCC) during Visit 3 or 4 (order counterbalanced).
  Interventions: Device: BrainSonix Pulsar 1002
- Sham LIFUP (Sham Comparator): All participants will receive sham modulation of the posterior cingulate cortex (PCC) during Visit 3 or 4 (order counterbalanced).
  Interventions: Device: BrainSonix Pulsar 1002

INTERVENTIONS:
Device: BrainSonix Pulsar 1002 — Device that delivers low intensity focused ultrasound

SUMMARY:
The specific aim of this proposed study is to investigate the feasibility and therapeutic potential of LIFUP in changing negative cognition in depression. Specifically, the investigators will study if modulating DMN activity can change maladaptive mind-wandering. The investigators hypothesize that DOWN-modulation of the posterior cingulate cortex (PCC), a key DMN node, will decrease DMN resting state functional connectivity, perfusion, and activation during a cognitive-affective task (description below). The investigators also hypothesize that DOWN-modulation of the PCC will be associated with decreased mind-wandering and increased mindfulness. Finally, the investigators hypothesize that the opposite will be true for UP-modulation of the PCC.

DETAILED DESCRIPTION:
The default mode network (DMN) is a network of structurally and functionally connected brain regions that was first identified during "passive" states. Since its initial discovery, the conceptualization of the DMN has evolved over time; the DMN has now been linked with a range of higher-order cognitive processes such as spontaneous, self-generated thoughts (i.e. mind-wandering) and thinking about oneself in the past, future, and in relation to others. Given the DMN's involvement in cognition, researchers have investigated its role in psychiatric disorders associated with cognitive issues, such as Major Depressive Disorder (MDD).

MDD is a mood disorder in which people experience a persistent negative mood or loss of interest or pleasure, thoughts of worthlessness and guilt, and/or suicidal ideation. The majority of literature suggests that currently depressed individuals have increased DMN resting-state functional connectivity at rest and greater DMN activation when processing negative stimuli. Researchers have suggested that this DMN hyperactivity reflects the tendency for depressed individuals to engage in negative cognition, such as maladaptive mind-wandering (i.e. task-irrelevant thought when individuals are supposed to be focused on a task) and rumination (i.e. negative, repetitive, self-focused thinking). Mind-wandering, in general, has been linked to unhappiness. Rumination is associated with the maintenance of a current depressive episode and is a predictor of future depressive episodes. Therefore, changing these forms of negative cognition, via modulation of DMN activity, could be of benefit to individuals with MDD.

One way of modulating DMN activity is to use brain stimulation. The investigators have previously used transcranial Direct Current Stimulation (tDCS) of a DMN brain region to effect a small yet significant reduction in mind-wandering behavior in a community sample. However, tDCS has low spatial specificity and neuroimaging was not used to determine if tDCS was actually changing mind-wandering via changes in DMN activity. Low Intensity Focused Ultrasound Pulsation (LIFUP) is a novel non-invasive brain stimulation method which has high spatial specificity, unlike other non-invasive brain stimulation methods such as Transcranial Magnetic Stimulation (TMS) and tDCS. Specifically, LIFUP can deliver acoustic energy to a brain region of a few millimeters in diameter. This method has been applied to the thalamus to restore consciousness to patients in minimally conscious states, and the investigators have been using this method in multiple IRB-approved studies as applied to the amygdala, ventral striatum, and entorhinal cortex.

Specific Aims:

The specific aim of this proposed study is to investigate the feasibility and therapeutic potential of LIFUP in changing negative cognition in depression. Specifically, the investigators will study if modulating DMN activity can change maladaptive mind-wandering. The investigators hypothesize that DOWN-modulation of the posterior cingulate cortex (PCC), a key DMN node, will decrease DMN resting state functional connectivity, perfusion, and activation during a cognitive-affective task (description below). The investigators also hypothesize that DOWN-modulation of the PCC will be associated with decreased mind-wandering and increased mindfulness. Finally, the investigators hypothesize that the opposite will be true for UP-modulation of the PCC.

Subject Selection:

Twenty participants (n = 40 healthy controls, n = 40 individuals with MDD) aged 18-64 years old will be recruited. The Structured Clinical Interview for DSM-5 Disorders, Research Version (SCID-5-RV)10 will be used to determine eligibility.

Subject Enrollment:

Participants will be recruited through email announcements at MGH, postings to college websites, and flyers (see attached flyer) posted at MGH and in the community (e.g., community centers, public libraries, coffee shops, restaurants, and laundromats). A phone screening will be performed to efficiently confirm likelihood that subjects will meet inclusion and exclusion criteria prior to committing time for further evaluation of eligibility.

Informed consent will be obtained prior to the performance of any protocol procedures. The informed consent document will be used to explain in simple terms the risks and benefits of study participation to the subject. The nature of the study will be fully explained to the subject by the PI, co-investigators or specially-trained study staff. The subject will be encouraged to ask questions pertaining to their participation in the study and the subject may take as much time as they feel necessary to consider his/her participation in the study as well as consult with family members or their physicians. Participation in this study is voluntary and the subjects may withdraw from the study at any time. The IRB-approved informed consent documents will be signed and dated by the subject and the person obtaining consent.

Study Procedures:

After providing study information and obtaining IRB approved informed consent, participants will complete up to five study visits on five different days.

Visit 1 (up to 1 hour):

For participants who are recruited as healthy controls, the SCID-5-RV will be administered to determine if the participant has no current or past history of any psychiatric disorders. For participants who are recruited as individuals with MDD, the SCID-5-RV will be administered to determine if the participant meets criteria for a current MDD diagnosis. Participants will be excluded from further study procedures if they do not meet the above-described criteria.

Visit 2 (up to 1 hour):

Participants will complete questionnaires assessing depressive symptoms, anxiety, mindfulness, and rumination.

After completing questionnaires, participants will practice the cognitive task they will be performing in the MRI scanner. Participants will complete a self-attribution task (Ghaznavi, Chou, Dougherty, & Nierenberg, 2023). Participants will see a series of trait adjectives and be asked to make a judgment about whether that personality trait applies to them (i.e. press a button indicating "Me" or "Not Me"). This task has been used by our lab to assess cognition and DMN activation in bipolar disorder.

After completing the practice computer task, participants will complete the MR Screening Safety form. After confirming the participant does not have MRI contraindications, they will be scanned using a 3 Tesla Siemens MRI scanner at the Athinoula A. Martinos Center for Biomedical Imaging. At baseline, we will collect a T1 MEMPRAGE structural scan, blood-oxygen-level-dependent (BOLD) resting state scan, Arterial Spin Labelled (ASL) scan, and a BOLD functional MRI scan paired with the task (described above). Participants will then exit the MRI scanner and will be asked to retrospectively report on their mind-wandering thoughts during the task. Participants will not receive LIFUP during this visit.

Visits 3 and 4 (up to 3.5 hours each; spaced 1 week apart):

At Visits 3 and 4, participants will complete the same questionnaires (described in Visit 2). To assess the subjective experience of LIFUP and its effects on mood, participants will rate their negative and positive mood on Visual Analog Scales as well as complete the 11-factor Altered States of Consciousness questionnaire (ASC) after LIFUP.

Participants will be scanned again with the same MRI sequences and complete the same computer task described in Visit 2, pre and post LIFUP.

LIFUP Sonication:

Participants will be fitted with the LIFUP device, the BX Pulsar 1002 (BrainSonix Corporation). The transducer will be placed on the head using landmarks and will be targeting the cluster in the PCC that was activated during the computer task in Visit 2. Participants will then receive either active or sham DOWN-modulation (Pulse Repetition Frequency = 10 Hz, Pulse-Width = 0.5 ms, Duty Cycle = 5%, ISPPA = 14.4 mW/cm2, 720 mW/cm2). The order will be counterbalanced across subjects. The sonications will be delivered in a 30-seconds on, 30-seconds off block design, for a total duration of 10 minutes. We are using the same LIFUP parameters in other IRB-approved LIFUP studies (IRB protocol #2019P000562 and IRB protocol #2019P001458) and these parameters have been safely used at other research collaborator sites at UCLA and MUSC. For sham sonication, a gel pad that absorbs ultrasound will be used with the transducer so that the ultrasound will not go through the skull and into the brain. For active sonication, a gel pad that allows the transmission of ultrasound waves will be used with the transducer. These gel pads look identical; this study will be double-blinded where study staff will not know which gel pad corresponded with active or sham LIFUP.

Visit 5 (up to 1 hour; spaced 1 week after Visit 4):

During this visit, participants will complete the same questionnaires (described in Visit 2).

Biostatistical Analysis:

fMRI data during the task will be analyzed using SPM12 software (Wellcome Department of Cognitive Neurology, London, UK). Individual subject-level data will be slice-time corrected, realigned and unwarped, coregistered to the individual's structural images, normalized, and smoothed. For LIFUP targeting, first-level contrast images will be created to identify BOLD activation in the PCC during self-judgments. To study the effects of LIFUP, first-level contrast images will be created comparing BOLD activation during the task before and after LIFUP. These contrast images will then be entered into a 2nd level random effects flexible factorial model. We will investigate whether there is a group (MDD versus healthy control) by condition (sham vs. active modulation) interaction on BOLD activation in DMN regions. Beta signal values will be extracted from DMN regions and we will investigate if there are significant correlations between DMN activation and our behavioral measures of depressive symptoms, anxiety, and mindfulness/mind-wandering.

BOLD resting state scan data will be similarly preprocessed and entered into CONN toolbox. The PCC will be used as a seed region and Fischer-transformed functional connectivity beta values with other DMN regions will be extracted for each individual subject. Repeated-measures ANOVAs will be conducted to again investigate whether there is a group by condition interaction on DMN resting state functional connectivity. Correlational analyses will also be performed to explore correlations with behavioral measures.

ASL data will be analyzed using Bayesian Inference for Arterial Spin Labeling MRI. Perfusion maps corresponding to pre and post LIFUP will be subtracted from each other to determine if there is decreased or increased perfusion in DMN regions associated with active modulation.

An updated statistical power analysis from our recent LIFUP study of the amygdala suggests that 40 participants will be necessary to achieve statistical significance (p < 0.05) in a voxel-based analysis. To increase our statistical power for comparing two groups, we will recruit 40 participants in each group (total n = 80).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age 18-64
3. Right-handed
4. Normal or corrected-to normal vision and hearing
5. For group with depression, current diagnosis of depression

Exclusion Criteria:

1. Active significant medical illness or neurological disorder
2. MRI scan contraindications (e.g., metal implant, claustrophobia, weigh over 250 pounds, etc.)
3. For healthy control group, any current or past history of psychiatric disorders

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Negative self-judgment frequency during task | 3 hours
  Changes in reported frequency of negative self-judgments during the self-attribution task before and after sham and active modulation
Default mode network activation during task | 3 hours
  Changes in Blood-Oxygen-Level Dependent activation in the default mode network during the self-attribution task before and after sham and active modulation
Rumination | 1 week
  Changes in Ruminative Responses Scale scores after the sham and active modulation sessions

SECONDARY OUTCOMES:
Depressive symptoms | 1 week
  Depressive symptoms as measured by the Beck Depression Inventory in the week after the active session
Default mode network connectivity | 3 hours
  Changes in default mode network resting state functional connectivity before and after sham and active modulation

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No